CLINICAL TRIAL: NCT04039620
Title: Sarcopenia in Acute Care Patients: Protocol for the European Collaboration of Geriatric Surveys: Sarcopenia 9+ European Academy for Medicine of Ageing (EAMA) Project
Brief Title: EAMA Sarcopenia in Acute Care Patients in 9+European Countries
Acronym: EAMA9+
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic and lack of funding necessary for continuation
Sponsor: Parc de Salut Mar (Other)
Collaborators: Jagiellonian University (Other); Université Libre de Bruxelles (Other); Agaplesion Bethesda Clinic Ulm, Ulm, Germany (Unknown); Slagelse Hospital (Other); Charles University, Czech Republic (Other); NOVA Medical School (Other); Karolinska Institutet (Other); Catholic University of the Sacred Heart (Other); University Hospital, Ghent (Other); University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/8355/I
Record Dates: First submitted 2019-03-06; First posted 2019-07-31 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Sarcopenia; Malnutrition
Keywords: Sarcopenia; Malnutrition; EWGSOP2; Older people; Acute care; Hospitalized
MeSH Terms: conditions — Sarcopenia; Malnutrition | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study, no interventions expected — No interventions are planned

SUMMARY:
This collaborative study in 9 geriatrics units across Europe aims to apply emerging research to clinical practice, following the "Action-Research Philosophy" (11). The overall goal is to improve care in patients with - and help prevent - sarcopenia. Understanding the frequency of and risk factors for developing sarcopenia in an acute hospital setting, may help shed light on potential interventions and thus inform the development of future therapeutic strategies. It involves crucial implications for research, clinical practice, and policy towards optimal aging.

DETAILED DESCRIPTION:
Background: Sarcopenia is a nutrition-related disease leading to physical impairment and adverse clinical outcomes. Data regarding its characteristics in hospitalized patients are limited.

Aim: This study will assess in older patients admitted to acute medical wards, the prevalence, incidence, and risk factors for development of sarcopenia, or alteration in its severity, and evaluate associated clinical adverse outcomes.

Methods: This collaboratively-designed, longitudinal prospective observational study will be carried out in patients aged >70 admitted to acute geriatric units in 9 European centers. The new sarcopenia diagnostic criteria of the European Working Group on Sarcopenia 2 (EWGSOP2) will be tested at admission and discharge, using isometric handgrip dynamometry, gait speed, and, pragmatically, calf circumference. There will be 3- and 12-month telephone follow-up (including the SARC-F questionnaire).

Discussion: Our study will be the first collaboration to assess the prevalence and incidence of sarcopenia (EWGSOP2) and its risk factors in hospitalized patients across Europe.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >70 admitted to acute hospital medical units

Exclusion Criteria:

* Length of hospital stay anticipated to be <24 hours
* Hip/lower limb fractures
* Major amputations of the lower leg
* Terminally ill patients admitted for palliative care

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients hospitalized in acute care units due to medical processes
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of sarcopenia as defined by the European consensus on definition and diagnosis (EWGSOP2) | One year (March 2019-March 2020)
  Prevalence sarcopenia in acute hospitalized older patients.
Incidence of sarcopenia as defined by the European consensus on definition and diagnosis (EWGSOP2) | One year (March 2019-March 2020)
  Incidence of sarcopenia in acute hospitalized older patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanchez Rodríguez, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Rodriguez D, Hope S, Piotrowicz K, Benoit F, Czesak J, Dallmeier D, Decker G, De Spiegeleer A, Hojmann AH, Hrnciarikova D, Marco E, Mendes D, Meza D, Nascimento P, Rodrigues A, Surquin M, Toscano-Rico M, Vankova H, Vetrano DL, Gasowski J, Van Den Noortgate N, Landi F. Sarcopenia in Acute Care Patients: Protocol for the European Collaboration of Geriatric Surveys: Sarcopenia 9+ EAMA Project. J Am Med Dir Assoc. 2019 Nov;20(11):e1-e3. doi: 10.1016/j.jamda.2019.04.030. Epub 2019 Jun 21. No abstract available. PMID 31230903
- See also: Sarcopenia in Acute Care Patients: Protocol for the European Collaboration of Geriatric Surveys: Sarcopenia 9+ EAMA Project. — http://www.ncbi.nlm.nih.gov/pubmed/31230903

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT04039620/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT04039620/ICF_001.pdf